CLINICAL TRIAL: NCT01904864
Title: A Single-center, Double-blinded, Randomized, 12 Week, Superiority Study in Infants and Young Children to Compare the Efficacy of NovaFerrum® Versus Ferrous Sulfate in the Treatment of Nutritional Iron Deficiency Anemia.
Brief Title: Comparison of NovaFerrum® vs Ferrous Sulfate Treatment in Young Children With Nutritional Iron Deficiency Anemia
Acronym: BESTIRON
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Gensavis Pharmaceuticals, LLC (Unknown)
Responsible Party: Principal Investigator, Patrick Leavey, Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FE15929
Record Dates: First submitted 2013-07-17; First posted 2013-07-22 (Estimated); Results first posted 2017-09-13 (Actual); Last update posted 2017-12-14 (Actual); Status verified 2017-11

CONDITIONS: Iron Deficiency Anemia
Keywords: randomized controlled trial; iron medication; Anemia; Hematologic Disease; Anemia, Iron deficiency; anemia, nutritional; ferrous sulfate; NovaFerrum®
MeSH Terms: conditions — Anemia, Iron-Deficiency; Anemia; Hematologic Diseases | interventions — ferrous sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NovaFerrum® (Active Comparator): Subjects randomized to this arm will receive a single daily dose (3mg/kg) of a 15 mg/ml elemental iron preparation, NovaFerrum®, for 12 weeks.
  Interventions: Drug: elemental iron (NovaFerrum®)
- Ferrous Sulfate (Active Comparator): Subjects randomized to this arm will receive a single daily dose (3mg/kg) of a 15 mg/ml elemental iron preparation, ferrous sulfate, for 12 weeks.
  Interventions: Drug: elemental iron (Ferrous Sulfate)

INTERVENTIONS:
Drug: elemental iron (NovaFerrum®) — single daily dose (3mg/kg) of a 15 mg/ml elemental iron preparation, NovaFerrum®, for 12 weeks
  Other Names: Generic Name: polysaccharide iron vitamin mineral complex
  Arms: NovaFerrum®
Drug: elemental iron (Ferrous Sulfate) — single daily dose (3mg/kg) of a 15 mg/ml elemental iron preparation, Ferrous Sulfate, for 12 weeks
  Other Names: Ferrous Sulfate
  Arms: Ferrous Sulfate

SUMMARY:
This study is a randomized, controlled, double-blinded single center trial to compare the efficacy of NovaFerrum® to ferrous sulfate for the treatment of nutritional iron deficiency anemia (IDA) in infants and young children.

Hypothesis: NovaFerrum® has greater efficacy than ferrous sulfate in increasing hemoglobin concentration during a twelve week course of treatment to subjects with iron deficiency anemia.

Primary Aim:

To compare the efficacy of NovaFerrum® to ferrous sulfate for the treatment of nutritional IDA in infants and young children as determined by increase in hemoglobin concentration.

Secondary Aims:

1. To compare the adverse effects of treatment for IDA between ferrous sulfate and NovaFerrum®
2. To compare normalization of iron stores as demonstrated by laboratory measures of IDA (ferritin, TIBC, reticulocyte hemoglobin content) between subjects treated with ferrous sulfate or NovaFerrum®
3. To compare the adherence to study medication between subjects on ferrous sulfate and NovaFerrum®
4. To demonstrate efficacy of a once daily dosing regimen in the treatment of nutritional IDA

DETAILED DESCRIPTION:
Screening/Baseline Assessment (Week 0):

* History and Physical Examination:
* Detailed history regarding medical disorders predisposing to iron deficiency and diet (breast feeding, iron fortified formula, cow's milk), including total daily amount.
* Review of existing medical records (including blood counts and iron studies) submitted by primary care provider or recorded on Children's electronic medical record.
* History of pica and/or other sequelae from iron deficiency.
* Details regarding prior or current iron oral therapy (dose, preparation, timing, response) or recent blood transfusions.
* Comprehensive physical exam (PE) (baseline visit) consisting of vital signs, general, HEENT, cardio-respiratory, abdominal, extremities and skin; Focused PE (Weeks 4 and 12) consisting of vital signs, general, cardio-respiratory, abdominal and skin.
* Laboratory (Only #3 below for research only, not standard of care):

  1. Complete blood count (CBC), reticulocyte count and reticulocyte hemoglobin content.
  2. Serum ferritin, iron and total body iron capacity (TIBC).

Treatment Interventions:

* Patients who meet eligibility criteria and whose parents provide written informed consent will be randomized in a 1:1 ratio to receive either ferrous sulfate drops (15 mg/ml) or NovaFerrum® drops (15 mg/ml).
* Subjects will be assigned to receive a single daily dose of 3 mg/kg elemental iron. Timing of study drug will be at bedtime.
* As a part of standard care, patients will be advised to reduce cow milk intake to a maximum 16 oz. daily and not to give any milk after medication administration. There will be no other dietary modification prescribed by the study.
* Other iron containing medications (including vitamins) will be discontinued.
* Families will be asked to make a daily diary entry documenting administration and adverse effects and return the diary at follow-up clinic visits.

Follow-up Phone Contact (Weeks 2, 6, 10 - not standard of care)

- Phone contact with parents will be made biweekly between scheduled visits (e.g. Weeks 2, 6, and 10) to assess adverse effects, promote strict adherence and remind them of the next scheduled visit.

Assessment During Follow-up Visits at Weeks 4, 8, and 12 after Initiation of Therapy (Follow-up visits during weeks 4 and 12 are standard of care; Follow-up visit at week 8 is for research only):

* Review of interval history and diet by direct questioning of the parents and review of diary regarding adherence, adverse effects of iron therapy (e.g., refusal to take, spitting/vomiting, abdominal pain, constipation, black stools, stained teeth). The diary will also contain distracter items to assess background "noise".
* Recording of other medications or intercurrent illnesses.
* Laboratory studies at each follow-up visit: CBC with red blood cell (RBC) indices, (MCV, RDW) reticulocyte count, reticulocyte hemoglobin content, serum ferritin, serum iron and total iron binding capacity.
* Blood lead measurement at week 4 (research only). Will repeated only if abnormal.
* Focused physical exam at 4 and 12 week visits

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 9 to < 48 months
2. IDA documented by hematologic indices (hemoglobin, MCV, RDW, reticulocyte count, reticulocyte hemoglobin content), serum ferritin, serum iron and total iron binding capacity

Exclusion Criteria:

1. Iron deficiency likely or definitely due to blood loss from the intestine or other sites.
2. Evidence of response to recent/current oral iron therapy, as determined by increase in hemoglobin by > 1.0 gm/dL and MCV by 5 fL above measurements prior to iron therapy
3. History or evidence of intestinal malabsorption
4. History of prior intravenous iron therapy
5. Major co-morbidity such as a serious chronic medical condition unrelated to iron deficiency apparent on history, physical examination, or laboratory tests
6. Other causes of anemia (sickle cell disease, thalassemia, other hemolytic anemia, bone marrow failure, etc.) apparent by history, physical examination, and/or laboratory tests.
7. High likelihood of suboptimal adherence by parents with study requirements (previous missed clinic visits)
8. Inability to tolerate oral medications
9. History of birth at < 30 weeks gestation
10. Other medical or social factors at discretion of treating physician

Ages: 9 Months to 48 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2013-07; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Leavey, MD, Principal Investigator — U Texas Southwestern
Locations (1):
- Children's Medical Center Dallas, Dallas, Texas, United States

REFERENCES:
- [Derived] Powers JM, Buchanan GR, Adix L, Zhang S, Gao A, McCavit TL. Effect of Low-Dose Ferrous Sulfate vs Iron Polysaccharide Complex on Hemoglobin Concentration in Young Children With Nutritional Iron-Deficiency Anemia: A Randomized Clinical Trial. JAMA. 2017 Jun 13;317(22):2297-2304. doi: 10.1001/jama.2017.6846. PMID 28609534

RESULTS

PARTICIPANT FLOW:
Groups:
- NovaFerrum® (Iron Polysaccharide Complex): Subjects randomized to this arm received a single daily dose (3mg/kg) of a 15 mg/ml elemental iron preparation of an iron polysaccharide complex (NovaFerrum®), for 12 weeks.
- Ferrous Sulfate: Subjects randomized to this arm received a single daily dose (3mg/kg) of a 15 mg/ml elemental iron preparation, ferrous sulfate, for 12 weeks.
Period: Overall Study
Arm/Group | NovaFerrum® (Iron Polysaccharide Complex) | Ferrous Sulfate
Started | 40 | 40
Completed | 31 | 28
Not Completed | 9 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NovaFerrum® (Iron Polysaccharide Complex) | Ferrous Sulfate | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Median (Full Range); unit: Months] | 23 [11 to 34] | 22 [10 to 37] | 23 [10 to 37]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 18 | 36
  Male | 22 | 22 | 44
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic white | 26 | 23 | 49
  Non-Hispanic white | 3 | 4 | 7
  Black | 4 | 5 | 9
  Asian | 2 | 2 | 4
  Native Hawaiian/Pacific Islander | 1 | 0 | 1
  >1 Race/ethnicity | 4 | 6 | 10
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40 | 40 | 80

OUTCOME MEASURES:

1. Primary Outcome: Hemoglobin Concentration Over Time
Description: The primary outcome will be the change in the peripheral blood hemoglobin concentration in grams/deciliter upon serial measurements at 0, 4, 8, and 12 weeks post-initiation of treatment. The primary analysis consists of a linear mixed regression model, which incorporates all subsequent time points into the model and includes treatment and time as covariates and patient random effects to account for correlation among longitudinal measurements from the same patients.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | NovaFerrum® (Iron Polysaccharide Complex) | Ferrous Sulfate
Number analyzed (Participants) | 40 | 40
g/dL
  Baseline | 7.7 (1.6) | 7.9 (1.5)
  4 Weeks | 9.3 (1.4) | 10.4 (1.3)
  8 Weeks | 10.5 (1.3) | 11.4 (1.3)
  12 Weeks | 11.1 (1.2) | 11.9 (1.2)
Statistical Analysis 1: Comparison: NovaFerrum® (Iron Polysaccharide Complex) vs Ferrous Sulfate; Test type: Superiority; p < 0.001, Regression, Linear; Mean Difference (Net) = 1.0, 95% CI 2-sided [0.4 to 1.6] — Change at 12 weeks compared

ADVERSE EVENTS:
Arm/Group | NovaFerrum® (Iron Polysaccharide Complex) | Ferrous Sulfate
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 1/40
Other Adverse Events (participants affected / at risk) | 32/40 | 29/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NovaFerrum® (Iron Polysaccharide Complex) (N=40) | Ferrous Sulfate (N=40)
Methemoglobinemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — One patient receiving ferrous sulfate experienced a transient episode of methemoglobinemia of unknown cause during week 4. The patient was successfully treated with methylene blue and continued in the study without recurrence.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NovaFerrum® (Iron Polysaccharide Complex) (N=40) | Ferrous Sulfate (N=40)
Gastrointestinal (Gastrointestinal disorders) | 32 (32) | 29 (29) — Patients reporting abdominal pain, vomiting, diarrhea, or constipation at any time point in the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No